CLINICAL TRIAL: NCT04955457
Title: BDNF Promoter Methylation: Effects on Cognition, Stress and Anxiety and Depression Symptom in Healthy Women.
Acronym: BDNFm
Status: Completed | Type: Observational
Sponsor: Ana Flávia Marçal Pessoa (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Sponsor-Investigator, Ana Flávia Marçal Pessoa, Co-investigator, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Other Study IDs: 3.159.669/2018
Record Dates: First submitted 2021-06-21; First posted 2021-07-08 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: BDNF; Memory Impairment; Stress; Well-being; Methylation
Keywords: BDNF methylation; Memory; women; Stress
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Healthy women active teachers — The neuropsychological testing data, psychometric measure, demographic, clinical and lifestyle information and blood samples were collected at similar time points. This group not received any intervention.

SUMMARY:
The purpose of this study is to explore the association between BDNF methylation and neurocognitive performance, perceived stress, and well-being in healthy women.

ELIGIBILITY:
Inclusion Criteria: (1)Brazilian female aged between 23 and 65 years and (2) currently working in the classroom

Exclusion Criteria:

1. diagnosis of depression
2. diagnosis of anxiety disorder
3. diagnosis of squizofrenia
4. report of an infectious condition in the last 15 days before collecting a blood sample;

Ages: 23 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female participants will be recruited from public schools linked to the "Diretoria Regional de Educação de Santo Amaro - DRESA" - a southern section of the São Paulo City Hall public education secretaryship.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Explore BDNF methylation level in healthy women active teachers | baseline
  Venous blood was obtained from all participants to DNA extraction and BDNF methylation analyses.
Explore episodic memory in healthy women active teachers | Baseline
  The RAVLT is a validated neuropsychologic test to evaluate learning and memory (episodic memory)an assessment of verbal learning over 5 trials and 30-minute delayed free recall
Explore working memory in healthy women active teachers | Baseline
  Investigates the capacity of working memory (auditory) and attention. It consists of two tables with different numbers, one with a direct order and another with a reverse order. The sequence of numbers is read aloud to the participant, one by one, where he must immediately repeat them to the examiner. The same happens with numbers in reverse order, but the participant must repeat the numbers backwards (reverse order). The maximum possible score to be reached in the forward order is 16 points, and in the reverse order 14 points totaling 30 points in the total score. For evaluation, the result must be compared with the standardization according to age.
Explore attention in healthy women active teachers | Baseline
  Trail Making Test (TMT): is used to assess divided attention, consisting of two parts (A and B). It also assesses motor function, mental flexibility, visual processing speed and aspects of sustained and alternating attention. In both parts, the participant must draw a path marked by numbers in the shortest time possible and without taking the pencil off the paper. In part A, you must draw a path marked by numbers in ascending order, from 1 to 25. Part B has a higher degree of difficulty, requiring greater cognitive demand from the participant, who must draw the path, now marked with numbers ranging from 1 to 13, alternating with letters, ranging from A to L, thus: 1-A-2-B-3-C... And so on. The score is measured by the total time the participant took to perform each task and compared with the standardization for their age group.
Explore selective attention in healthy women active teachers | Baseline
  • Stroop Test: Allows you to detect neurological and brain problems and is also used to check and measure levels of concentration and cognitive functions, selective attention and speed of processing information. The test must be applied to adults over 25 years of age and consists of three tasks: the first in reading words, the second in naming colors, and the third in identifying and naming the color of each word that is written in distinct colors from its nomenclature, which is called the interference effect (or stroop effect). The score is obtained by scoring total correct answers in each of these tasks, and compared with the current standardization.
Explore perceived stress in healthy women active teachers | Baseline
  Perceived Stress Scale (PSS): is used to assess the individual's perception of stress (subjective stress assessment), where it should be noted how uncontrollable and unpredictable the events of their life experienced in the last month seem to be. The test consists of 10 items, 6 of positive aspects and 4 of negative aspects, and must be answered within a Likert-type frequency scale (ranging from 0 - Never to 4-Always). For its evaluation, all the answers must be added together to obtain a total perceived stress score, which must be compared with the standardization of the test for the equivalent population
Explore resilience in healthy women active teachers | Baseline
  • Connor-Davidson Resilience Scale (CD-RISC): a 25-item scale divided into 5 factors, namely: personal competence, confidence in one's instincts, positive acceptance of change, tolerance in the face of adversity, control and spirituality. The scale is self-applicable and the participant must mark answers ranging from 0 (never true) to 4 (always true). The result is obtained through the sum of the total score, which can range from 0 to 40 points, where the higher the score, the greater the participant's degree of resilience.
Explore psychological well-being in healthy women active teachers | Baseline
  • Psychological Well-Being Scale (PWBS): the scale consists of 84 items, subdivided into 6 scales that assess the dimensions of psychological well-being, with 14 items each. The answers are obtained through a Likert-type scale, ranging from 0 (totally disagree) to 6 (totally agree). The subscales are divided as follows: Self-acceptance, Positive relationship with others, autonomy, mastery of the environment, purpose in life and personal growth. The result is obtained through the sum of the items of each subscale, and the higher the score, the better the levels of psychological well-being according to each subscale.
Explore positive and negative affect in healthy women active teachers | Baseline
  • Positive and negative affect scale (PANAS): Aims to identify the dimensions of affect of subjective well-being, through 20 items provided, where participants must indicate how they have been feeling lately. These items are distributed into 10 of subjective emotions that comprise negative affects, and 10 items that comprise positive affects, being issued on a 5-point Likert scale ranging from 1 (not at all) to 5 (extremely).
Explore anxiety and depression symptoms in healthy women active teachers | Baseline
  • Hospital Anxiety and Depression Scale (HADS): It was developed to identify probable and possible levels and cases of Anxiety and Depression in clinical and non-clinical populations. It consists of 14 items divided into two subscales of 7 items each, where one comprises questions to identify signs of anxiety disorders, and the other of depression. The answers range from 0 to 3 points, ranging from absent to very frequent, with a maximum score of 21 points. The cutoff point obtained in the literature for both subscales is ≥ 9 points

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Rodrigues de Oliveira, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, WI, Brazil